CLINICAL TRIAL: NCT06332742
Title: Real-world Evaluation of the Clinical Efficacy of Qingxin Zishen Decoction in Patients With Reduced Ovarian Reserve
Brief Title: Real-world Evaluation of Qingxin Zishen Decoction on Ovarian Reserve Function Clinical Efficacy in Patients With Decreased
Status: Recruiting | Type: Observational
Sponsor: Yun Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Chen, chief physician, Jiangsu Province Hospital of Traditional Chinese Medicine
Organization: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Other Study IDs: QXZS for DOR
Record Dates: First submitted 2024-03-03; First posted 2024-03-27 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Decreased Ovarian Reserve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposome group: 5g lotus seed heart, 3g coptis, 15g uncaria, 15g fried jujube kernel, 10g dried rehmannia glutinosa, 9g dogwood meat, 10g salvia miltiorrhiza, 30g floating wheat.
  1 dose per day, decocted in water twice, 200ml each time, taken warmly after breakfast and dinner
- Non-exposed group: All patients who met the inclusion criteria and did not use Qingxin Zishen Decoction.

SUMMARY:
A prospective cohort study evaluated the clinical efficacy of Qingxin Zishen Decoction

ELIGIBILITY:
1.AMH AMH <1.1ng/ml 2.AFC: AFC <5~7 ovaries on both sides 3.Basic FSH: Basal FSH for two consecutive menstrual cycles ≥10 IU/L 4.Aged between 25 and 45 years old, female.

1. Those with reduced ovarian function caused by ovarian or uterine surgery, radiotherapy and chemotherapy;
2. Liver function (AST or ALT) and renal function (BUN or Ccr) are greater than 2 times the normal value;
3. Patients with a history of mental illness or legal disability
4. Those who have used endocrine-affecting drugs within 3 months before the study, estrogen, progesterone or related compound preparations, oral contraceptive pills, Chinese medicines or Chinese patent medicines related to the treatment of premature ovarian failure. Our hospital's preparations include Wu Turtle Rejuvenation Oral Liquid and Kuntai Capsules.
5. Patients with unexplained irregular vaginal bleeding
6. Patients who are participating in clinical trials of other drugs
7. For women who want to have children, those whose spouse's semen test fails to meet the standard will be excluded.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 1. Those who meet the diagnostic criteria for hypoovarian reserve disease and the TCM syndrome differentiation criteria for heart and kidney disharmony.
  2. Aged between 25 and 45 years old, female.
  3. Informed consent and voluntary participation.
  4. The process of obtaining informed consent should comply with GCP regulations.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Traditional Chinese medicine syndrome score | Keep truthful case records and medication records for patient during the initial diagnosis, 3rd month, 6th month and 12th month of treatment
  Traditional Chinese medicine syndrome score
serum sex hormone levels | Keep truthful case records and medication records for patient during the initial diagnosis, 3rd month, 6th month and 12th month of treatment
  SHBG stands for sex hormone binding globulin. It's a protein made mostly in your liver. It binds (attaches) to sex hormones in your blood.
serum AMH levels | Keep truthful case records and medication records for patient during the initial diagnosis, 3rd month, 6th month and 12th month of treatment
  An AMH test measures levels of anti-mullerian hormone, which corresponds to a person's egg count.
transluminal ultrasound evaluation of ovarian antral follicles and other parameters (AFC) | Keep truthful case records and medication records for patient during the initial diagnosis, 3rd month, 6th month and 12th month of treatment
  Antral follicle count is rightly done on day 3 of the cycle by a Trans vaginal ultrasound. Initially the ovarian volume of both the ovaries is calculated.

SECONDARY OUTCOMES:
Seven items of thyroid function | Keep truthful case records and medication records for patient during the initial diagnosis, 3rd month, 6th month and 12th month of treatment
  The thyroid gland produces hormones that regulate the body's metabolic rate, growth and development. It plays a role in controlling heart, muscle and digestive function, brain development and bone maintenance.
natural pregnancy rate | Keep truthful case records and medication records for patient during the initial diagnosis, 3rd month, 6th month and 12th month of treatment
  A woman in her early to mid-20s has a 25-30% chance of getting pregnant every month. Fertility generally starts to slowly decline when a woman is in her early 30s, and after the age of 35 the decline speeds up. By age 40, the chance of getting pregnant in any monthly cycle is around 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Hospital of Traditional Chinese Medicine Affiliated to Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No